CLINICAL TRIAL: NCT04096781
Title: Engaging Patients to Help Achieve Increased Patient Choice and Engagement for AFib Stroke Prevention
Acronym: ENHANCE-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: American Heart Association (Other); East Carolina University (Other); Ochsner Health System (Other); The Cleveland Clinic (Other); The Cooper Health System (Other)
Responsible Party: Principal Investigator, Paul Wang, Professor of Medicine (Cardiovascular Medicine), Stanford University Medical Center, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 50864
Record Dates: First submitted 2019-09-09; First posted 2019-09-20 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Atrial Fibrillation; Atrial Flutter; Stroke; Cardiac; Heart Failure; Arrhythmia
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter; Stroke; Heart Failure; Arrhythmias, Cardiac

STUDY DESIGN:
Intervention Model Description: A Shared Decision-Making pathway focused on a digital shared decision-making tool (SDMT) that is augmented by a clinician tool and an optional lay coach
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shared Decision Making Tool (SDMT) (Experimental)
  Interventions: Behavioral: SDMT
- Usual Care (Active Comparator)
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: SDMT — The intervention involves a clear pathway centered on the use of a web-based decision tool. This tool aims to support the shared decision-making process for anticoagulation for stroke prevention in atrial fibrillation. This web-based tool will be used both by the participants as well the physician responsible for atrial fibrillation decision making.
  Arms: Shared Decision Making Tool (SDMT)
Behavioral: Usual Care — The participants will receive usual care.
  Arms: Usual Care

SUMMARY:
A multi-center, randomized controlled 2-arm trial comparing the effectiveness of an innovative shared decision-making pathway and usual care for Atrial Fibrillation Stroke Prevention

DETAILED DESCRIPTION:
This study will test to see if a new type of decision-making process tool, called a Shared Decision Making Pathway, can make a difference in decreasing the risk of stroke due to a condition called Atrial Fibrillation (AFib.) This online tool is designed to help doctors and patients decide together on treatment options for AFib.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 y/o
* Non-valvular atrial fibrillation or atrial flutter (AFib)
* CHA2DS2-VASc stroke score of:

  * Men: 1 or more
  * Women: 2 or more
* Able to consent in English or Spanish (if resources allow) and follow study instructions

Exclusion Criteria:

* Moderate to severe mitral stenosis
* Mechanical valve replacement
* Absolute contraindication to anticoagulation (Based on clinician judgment)
* Indication for anticoagulation therapy for a condition other than atrial fibrillation
* Left atrial appendage exclusion (by surgery or device placement)
* At the clinical discretion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1001 (Actual)
Dates: Start 2019-12-18 (Actual); Primary Completion 2022-06-23 (Actual); Study Completion 2022-08-17 (Actual)

PRIMARY OUTCOMES:
Decisional Conflict Scale | Visit 2 (1-month follow-up)
  The Decisional Conflict Scale is a 16 Item scale on whether the participants have enough information to make a clear decision. Each item scored from 1-5, where 1 indicates clarity and 5 indicates confusion, with total score ranging from 16-80

SECONDARY OUTCOMES:
Decisional Conflict Scale (16 items) | Visit 1 (Post Clinic Visit), Visit 2 (1-month follow up), Visit 3 (6-month follow-up)
  The Decisional Conflict Scale is a 16 Item scale on whether the participants have enough information to make a clear decision. Each item scored from 1-5, where 1 indicates clarity and 5 indicates confusion, with total score ranging from 16-80
Decision Regret Scale (5 items) | Visit 1 (Post Clinic Visit), Visit 2 (1-month follow up), Visit 3 (6-month follow-up)
  Decision Regret Scale, is scored from 1-5, where 1 indicates they made the right decision and 5 indicates they made the wrong decision. This scale ranges from 5-25
Weighted composite outcome scale according to patient preference | Visit 1 (Post Clinic Visit), Visit 2 (1-month follow up), Visit 3 (6-month follow-up)
  Patient-selected weighted composite outcome scale is a composite scale to consider both decisional conflict and decisional regret scales simultaneously according to the priority based on the survey of 100 potential participants. The rationale for this endpoint is to consider not only the preference of majority patients (73%) but also the minority (27%) participants who prefer the decisional regret scale
Preparation for Decision Making Scale (10 items) | Visit 1 (Post Clinic Visit), Visit 2 (1-month follow up), Visit 3 (6-month follow-up)
  Preparation for Decision Making scale assesses a patient's perception of how useful a decision aid or other decision support intervention is in preparing the respondent to communicate with their practitioner at a consultation focused on making a health decision
Utah-Stanford Atrial Fibrillation Knowledge Assessment | Baseline, Visit 1 (Post Clinic Visit), Visit 2 (1-month follow up), Visit 3 (6-month follow-up)
  Newly developed assessment for this study to record Atrial Fibrillation Knowledge
Quality of Communication (Based on CAHPS Clinician & Group Survey) | Visit 1 (Post Clinic Visit)
  CAHPS 3-item modified version
Atrial Fibrillation Severity Scale (AFSS) | Baseline, Visit 2 (1-month follow up), Visit 3(6-month follow-up)
  The University of Toronto Atrial Fibrillation Severity Scale (AFSS) is a questionnaire designed for patients with AFib. It consists of 19 items combined into 3 parts to capture total AF burden, health care utilization, and the severity of AFib related symptoms
Collaborative Agreement on Decision | Visit 1 (Post Clinic Visit)
  Assess the collaborative agreement (1. Patient Reported Outcome 2) Clinician Reported
Clinician Satisfaction of the Decision Aid: Physician Survey | Visit 1 (Post Clinic Visit)
  Clinician Satisfaction of the Decision Aid as assessed by a physician survey on shared decision making
Patient Satisfaction of the Decision Aid: Patient Survey | Visit 1 (Post Clinic Visit)
  Patient Satisfaction of the Decision Aid as assessed by Patient survey on shared decision making
Length of Visit at visit 1 (clinician) | Visit 1 (Post Clinic Visit)
  Compare treatment arm on the length of visit
Anticoagulant Choice (Patient follow up questions on Anticoagulant use) | Visit 1 (Post Clinic Visit), Visit 2 (1-month follow up), Visit 3 (6-month follow-up)
  Decision on anticoagulation choice as assessed by patient follow up questions
Anticoagulation Persistence and adherence (Patient follow up questions on Anticoagulant use) | Visit 2 (1-month follow up), Visit 3 (6-month follow-up)
  Persistence and adherence to anticoagulation among participants selecting anticoagulation, as assessed by Patient follow up questions
Stroke or TIA or Deep Venous Thrombosis or Pulmonary Embolus | Visit 2 (1-month follow up), Visit 3 (6-month follow-up), Unscheduled
  Incidence of Stroke or TIA or Deep Venous Thrombosis or Pulmonary Embolus
Death | Visit 2 (1-month follow up), Visit 3 (6-month follow-up), Unscheduled
  Incidence of Death

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Wang, MD, Principal Investigator — Stanford University; Randall S Stafford, MD, Principal Investigator — Stanford University
Locations (5):
- United States (5):
  - Stanford University, Palo Alto, California
  - Ochsner Medical Center, New Orleans, Louisiana
  - Cooper University Hospital, Camden, New Jersey
  - East Carolina University, Greenville, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baykaner T, Pundi K, Lin B, Lu Y, DeSutter K, Lhamo K, Garay G, Nunes JC, Morin DP, Sears SF, Chung MK, Paasche-Orlow MK, Sanders LM, Bunch TJ, Hills MT, Mahaffey KW, Stafford RS, Wang PJ. The ENHANCE-AF clinical trial to evaluate an atrial fibrillation shared decision-making pathway: Rationale and study design. Am Heart J. 2022 May;247:68-75. doi: 10.1016/j.ahj.2022.01.013. Epub 2022 Jan 28. PMID 35092723
- [Background] Nunes JC, Baykaner T, Pundi K, DeSutter K, True Hills M, Mahaffey KW, Sears SF, Morin DP, Lin B, Wang PJ, Stafford RS. Design and development of a digital shared decision-making tool for stroke prevention in atrial fibrillation. JAMIA Open. 2023 Feb 2;6(1):ooad003. doi: 10.1093/jamiaopen/ooad003. eCollection 2023 Apr. PMID 36751465
- [Background] Chung MK, Fagerlin A, Wang PJ, Ajayi TB, Allen LA, Baykaner T, Benjamin EJ, Branda M, Cavanaugh KL, Chen LY, Crossley GH, Delaney RK, Eckhardt LL, Grady KL, Hargraves IG, True Hills M, Kalscheur MM, Kramer DB, Kunneman M, Lampert R, Langford AT, Lewis KB, Lu Y, Mandrola JM, Martinez K, Matlock DD, McCarthy SR, Montori VM, Noseworthy PA, Orland KM, Ozanne E, Passman R, Pundi K, Roden DM, Saarel EV, Schmidt MM, Sears SF, Stacey D, Stafford RS, Steinberg BA, Youn Wass S, Wright JM. Shared Decision Making in Cardiac Electrophysiology Procedures and Arrhythmia Management. Circ Arrhythm Electrophysiol. 2021 Dec;14(12):e007958. doi: 10.1161/CIRCEP.121.007958. Epub 2021 Dec 6. PMID 34865518
- [Background] Pundi K, Baykaner T, True Hills M, Lin B, Morin DP, Sears SF, Wang PJ, Stafford RS. Blood Thinners for Atrial Fibrillation Stroke Prevention. Circ Arrhythm Electrophysiol. 2021 Jun;14(6):e009389. doi: 10.1161/CIRCEP.120.009389. Epub 2021 Jun 11. No abstract available. PMID 34111936
- [Background] Ajayi TB, Remein CD, Stafford RS, Fagerlin A, Chung MK, Childs E, Benjamin EJ. Cross-Center Virtual Education Fellowship Program for Early-Career Researchers in Atrial Fibrillation. Circ Arrhythm Electrophysiol. 2020 Nov;13(11):e008552. doi: 10.1161/CIRCEP.120.008552. Epub 2020 Oct 8. PMID 33031707
- [Background] Nunes, J.C., Shah, S., Fazal, M. et al. Patient Education Strategies to Improve Risk of Stroke in Patients with Atrial Fibrillation. Curr Cardiovasc Risk Rep 16, 249-258 (2022). https://doi.org/10.1007/s12170-022-00709-8.
- [Background] Pourshams I, Lin B, Wang PJ, Stafford RS. Decision-Making Experiences and Decisional Regret in Patients Receiving Implanted Cardioverter-Defibrillators. Heart Mind 2022; 6(1): 32-5. doi: 10.4103/hm.hm_51_21
- [Result] Wang PJ, Lu Y, Mahaffey KW, Lin A, Morin DP, Sears SF, Chung MK, Russo AM, Lin B, Piccini J, Hills MT, Berube C, Pundi K, Baykaner T, Garay G, Lhamo K, Rice E, Pourshams IA, Shah R, Newswanger P, DeSutter K, Nunes JC, Albert MA, Schulman KA, Heidenreich PA, Bunch TJ, Sanders LM, Turakhia M, Verghese A, Stafford RS. Randomized Clinical Trial to Evaluate an Atrial Fibrillation Stroke Prevention Shared Decision-Making Pathway. J Am Heart Assoc. 2023 Feb 7;12(3):e028562. doi: 10.1161/JAHA.122.028562. Epub 2023 Feb 7. PMID 36342828